CLINICAL TRIAL: NCT03946761
Title: Evaluation of Fluorescence Imaging in Hepatobiliary Surgery
Brief Title: Fluorescence Imaging in Hepatobiliary Surgery
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: One of the main investigators is leaving the University.
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 201904180
Record Dates: First submitted 2019-04-30; First posted 2019-05-13 (Actual); Last update posted 2022-01-24 (Actual); Status verified 2022-01

CONDITIONS: Hepatobiliary Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Cancer goggle system (Experimental): * The surgical procedure will be performed according to standard practice, with the exception of microdosing of ICG & visualization of biliary/liver anatomy using the cancer goggles system
  * The surgeon will start with a peripherally injected microdose of 0.02 mg of ICG & will inject an additional 0.02mg every 5 minutes until a noticeable fluorescent change in the liver is observed. If a change is not observed after 0.14 mg has been injected then the microdosing regimen will stop. Output video from the cancer goggles will be recorded and saved for post-surgical analysis.
  * Following resection of the liver parenchyma, the portal area and the cut surface of the liver will be analyzed for the identification of bile ducts leaks with or without cancer goggles.
  Interventions: Device: Cancer goggle system

INTERVENTIONS:
Device: Cancer goggle system — -The cancer goggle system is being used as a non-significant risk device

SUMMARY:
A current gap in the use indocyanine green fluorescence to isolate the biliary system is the dosing amount necessary to fluoresce the biliary system without "over" fluorescing the liver and gallbladder. Over fluorescing surrounding structures such as the liver and gallbladder saturates the image and makes it impossible to identify biliary leaks or differentiate branches of the common bile duct using fluorescent imaging devices. The over dosing does not affect the standard of care procedure, but eliminates the added benefit of the fluorescent imaging technology. The use of "microdoses" (approximately 0.1 mg) of indocyanine green has been trialed and shown promise in some patients. This study aims to do an in depth study utilizing the Cancer goggle systems fluorescent imaging system to determine the correct dose needed to isolate the biliary system without over fluorescing surrounding structures. This dosing study could additionally serve as a pilot study for follow on research using indocyanine green and fluorescent imaging in hepatobiliary surgery.

ELIGIBILITY:
Inclusion Criteria:

* Planned open liver resection or ablation.
* At least 18 years of age.
* Able to understand and willing to sign a written informed consent document.

Exclusion Criteria:

-History of allergic reactions attributed to ICG, iodine, iodine dye, or other agents used in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-12-31 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
The minimum dose of the ICG that causes initial fluorescence of the liver | Through completion of surgery for all participants enrolled (estimated to take 1 year)

SECONDARY OUTCOMES:
The visible status of the bile ducts and/or bile leaks from the cut surface of the liver at ICG doses administered in our dosing regimen | Through completion of surgery for all participants enrolled (estimated to take 1 year)

CONTACTS AND LOCATIONS:
Overall Officials: Chet Hammill, M.D., FACS, Principal Investigator — Washington University School of Medicine

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu